CLINICAL TRIAL: NCT00545987
Title: Evaluation of Local and Systemic Reactogenicity Following Serial Administration of ADVAX, a Clade C DNA Vaccine, ADVAX e/g + ADVAX p/N-t, by Ichor TriGrid™ in Vivo Electroporation to HIV-Uninfected, Healthy Volunteers
Brief Title: Study of a Potential Preventive Vaccine Against HIV in Healthy Volunteers
Acronym: ADVAX-EP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Aaron Diamond AIDS Research Center (Other); Bill and Melinda Gates Foundation (Other); Ichor Medical Systems Incorporated (Industry); International AIDS Vaccine Initiative (Network)
Responsible Party: David Ho, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DHO-0614
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infections
Keywords: HIV vaccine; HIV; AIDS; prevention; HIV/AIDS; HIV Preventative Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intramuscular injection (Active Comparator): administration of an HIV-1 vaccine by conventional intramuscular injection
  Interventions: Device: conventional intramuscular injection
- TriGrid Delivery System (Experimental): electroporation-mediated intramuscular delivery using the TriGridTM device by Ichor Medical Systems, Inc.
  Interventions: Device: TriGrid™ Delivery System

INTERVENTIONS:
Device: TriGrid™ Delivery System — Subjects will be administered the study drug using Ichor Medical Systems' intramuscular TriGrid™ delivery device.
  Arms: TriGrid Delivery System
Device: conventional intramuscular injection — administration of an HIV-1 vaccine encoding the gag, env, pol, nef, and tat antigens (ADVAX)by conventional intramuscular injection
  Arms: intramuscular injection

SUMMARY:
This study will test the safety of a HIV DNA vaccine after it is injected into your muscle using an electroporation device (TriGrid™ Delivery System made by Ichor Medical Systems), and will test the ability of the vaccine to help your body make antibodies and T-Cells.

In this study, we would like to learn about the effects that electroporation of the HIV DNA has on you and your immune system.

DETAILED DESCRIPTION:
Over 40 million people worldwide are currently infected with HIV, the virus that causes AIDS (Acquired Immune Deficiency Syndrome). The number of new cases continues to rise at an alarming rate. Other infectious diseases, such as smallpox or poliomyelitis, have been controlled, or even eliminated, by vaccination programs. Many experts believe that an HIV vaccine offers the best hope for controlling the epidemic.

Many different possible HIV vaccines are currently being developed and tested.

The ADVAX vaccine which you will receive is one vaccine that has been tested. To date, one to three doses of the ADVAX vaccine have been given to 45 individuals in a study that took place between December 2003 and October 2005 at the Rockefeller University and the University of Rochester and it appears to be safe. The difference between this ADVAX study and the previous one is that you will only receive two doses of the vaccine or placebo by either standard intramuscular injection or by "electroporation."

This study is part of a broader research effort to see if changes in the way vaccines are given can make vaccines more effective.

The results of other studies suggest that using regular needles may not be the most potent way to inject this type of vaccine. This is why we are studying a new method of injection called electroporation.

Electroporation uses a device that injects substances into muscle along with small amounts of electricity. This device has been used to a limited extent in human subjects and has been shown to be more effective than regular needles and safe when tested in animals. Devices similar to this have been used in many studies to deliver chemotherapy directly into patients' tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Men and Women
2. Ages 18 to 60
3. Not considered to be at high risk to acquire HIV infection.

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically significant abnormality on history or examination
3. Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
4. Hepatitis B; hepatitis C
5. Syphilis
6. If female, pregnant, planning a pregnancy during the trial period, or breastfeeding
7. Receipt of a live attenuated vaccine (other than influenza) within 30 days or other vaccine within 14 days of ADVAX vaccination
8. Receipt of blood transfusion or blood products 6 months prior to vaccination
9. Participation in another clinical study of an investigational product currently or within past 3 months, or expected participation while enrolled in this study
10. History of severe local or systemic reactogenicity to vaccination or history of severe allergic reactions
11. Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicidal attempt or ideation in the previous 3 years
12. Any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators
13. Individuals in which a skin-fold measurement of the cutaneous and subcutaneous tissue for all eligible injection sites (deltoid muscles with intact lymph drainage) exceeds 40 mm
14. In the opinion of the investigator, unlikely to comply with protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of an intramuscular prime and boost injection of the ADVAX DNA-based HIV vaccine via TriGrid™ electroporation at all three dosing levels | wk. 1,2, 4, 9, 10, 12, 16, 24, 36, 48 and 56

SECONDARY OUTCOMES:
• To evaluate the immunogenicity of an intramuscular prime and boost injection of the ADVAX DNA-based HIV vaccine via TriGrid™ electroporation compared to placebo or standard syringe injection at all three dosing levels. | wk. 1,2, 4, 9, 10, 12, 16, 24, 36, 48 and 56

CONTACTS AND LOCATIONS:
Overall Officials: David Ho, M.D., Principal Investigator — The Aaron Diamond AIDS Research Center
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Vasan S, Hurley A, Schlesinger SJ, Hannaman D, Gardiner DF, Dugin DP, Boente-Carrera M, Vittorino R, Caskey M, Andersen J, Huang Y, Cox JH, Tarragona-Fiol T, Gill DK, Cheeseman H, Clark L, Dally L, Smith C, Schmidt C, Park HH, Kopycinski JT, Gilmour J, Fast P, Bernard R, Ho DD. In vivo electroporation enhances the immunogenicity of an HIV-1 DNA vaccine candidate in healthy volunteers. PLoS One. 2011;6(5):e19252. doi: 10.1371/journal.pone.0019252. Epub 2011 May 16. PMID 21603651
- See also: The Aaron Diamond AIDS Research Center — http://www.adarc.org/